CLINICAL TRIAL: NCT00031135
Title: Prevention of TPN-Associated Hepatic Steatosis: A Placebo Controlled Trial
Brief Title: Total Parenteral Nutrition-Associated Liver Disease
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Northwestern University (Other)
Organization: FDA Office of Orphan Products Development (U.S. Federal Agency)
Allocation: Randomized | Masking: Double | Purpose: Prevention
Other Study IDs: FD-R-1994-01; FD-R-001994-01
Record Dates: First submitted 2002-02-26; First posted 2002-02-27 (Estimated); Last update posted 2015-03-25 (Estimated); Status verified 2002-01

CONDITIONS: Liver Diseases
Keywords: Parenteral Nutrition, Total; Lipotropic Agents; Choline
MeSH Terms: conditions — Liver Diseases; Hyperphagia | interventions — Choline

INTERVENTIONS:
Drug: Choline Chloride

SUMMARY:
This is a study to determine whether choline, when added to total parenteral nutrition (TPN), can help prevent the development of hepatic steatosis, a liver disease, in patients on TPN.

DETAILED DESCRIPTION:
Choline deficiency-induced hepatic steatosis occurs in patients that require long-term TPN and may progress to significant hepatic disease and death. Initial studies indicate choline-supplemented TPN may reverse TPN-associated hepatic steatosis.

Choline chloride or placebo will be added to each patient's TPN for 16 weeks by the hospital or pharmacy providing their usual TPN. Patients will receive their TPN in the hospital until they are medically stable for discharge. If patients are discharged before study completion, the pharmacy will deliver the TPN supply to them. Evaluation of hepatic steatosis is done by CT scans and blood analyses. Blood will be drawn on a biweekly basis during the first 4 weeks and at Week 8, 12, 16 or withdrawal. CT scans will be done at Week 4, 8, 16, or withdrawal.

Completion date provided represents the completion date of the grant per OOPD records

ELIGIBILITY:
Inclusion criteria:

* Underlying pathology may include, but is not limited to: short bowel syndrome, chronic pancreatitis, pancreatic pseudocysts, pseudo-obstruction, enterocutaneous fistula, entero-enteric fistula, or malabsorption syndrome.
* Requirement for TPN to supply greater than 85 percent of nutritional needs for at least 16 weeks.

Exclusion criteria:

* Not receiving lipid emulsion with TPN regimen
* Albumin less than 2.5 g/L
* Renal failure requiring hemo- or peritoneal dialysis
* Hepatic failure (PT greater than 2 times control)
* Diabetes
* Hepatitis C
* AIDS
* Concurrent hospitalization for organ transplantation or rejection treatment
* Concurrent cholinergic medication
* Positive pregnancy test
* Refusal to use an acceptable method of birth control
* Ethanol abuse
* More than 40 kcal/kg/day ideal body weight
* Obesity with ensuing weight loss
* Use of IV tetracycline, valproic acid, corticosteroids, methotrexate, or amiodarone

Ages: 21 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2001-09; Study Completion 2005-09

CONTACTS AND LOCATIONS:
Locations (1):
- Northwestern University, Chicago, Illinois, United States